CLINICAL TRIAL: NCT06248632
Title: Effect of Burosumab on the Inflammatory Profile of Patients With X-linked Hypophosphatemic Rickets FLAM-XLH
Acronym: FLAM-XLH
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1216
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: X-Linked Hypophosphatemic Rickets
Keywords: XLH; Burosumab; inflammation
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Inflammation | interventions — Interleukin-6; Interleukin-8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with genetically confirmed XLH diagnosis treated with bursosumab: Blood sampling at D0 and D7 for monocytic cell extraction in vitro
  Interventions: Other: Expression of inflammatory markers (Il6, Il8, Il1β, CXCL1, CCL2, CXCR3, Il1R, Il6R)

INTERVENTIONS:
Other: Expression of inflammatory markers (Il6, Il8, Il1β, CXCL1, CCL2, CXCR3, Il1R, Il6R) — Expression of inflammatory markers obtained from circulating monocytic cells of XLH

SUMMARY:
X-linked hypophosphataemia (XLH) is a rare genetic disorder associated with increased circulating levels of the hormone FGF23, most commonly through mutation of the PHEX gene. XLH is associated with a wide range of clinical manifestations in children and adults, all of which can impact on their health-related quality of life.

Conventional treatment (or standard of care, SOC) consists of phosphate supplementation and active vitamin D analogues. The management of patients with XLH has been modified in France since 2018 with the authorisation of the anti-FGF23 antibody, burosumab, in paediatrics (and in 2020 in adults).

A propensity for overweight/obesity has recently been demonstrated in these patients. Could extra-skeletal effects of FGF23, in particular on the inflammatory profile of patients, be responsible for these manifestations? Obesity has been associated with inflammation in other populations. In terms of inflammation, there is a close link between FGF23 and inflammation: inflammatory cytokines increase the production of FGF23, which in turn increases inflammation by stimulating the production of inflammatory cytokines. Osteoclastogenesis and inflammation are linked and inflammation has been shown to increase bone resorption.

In a recent study, the investigators showed that osteoclastogenesis was significantly impaired in cells obtained from XLH patients compared with control patients, and that osteoclasts obtained from XLH children showed higher gene expression of inflammatory markers than controls. Interestingly, no difference was observed in circulating monocytic cells between the two patient subgroups, conservative treatment and burosumab, whereas the inflammatory profile at the end of osteoclastic differentiation was reduced in cells derived from patients receiving burosumab.

The aim of this study is therefore to investigate the inflammatory profile of circulating monocytic cells on the day of burosumab injection (D0) and seven days later (peak effect of anti-FGF23).

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with genetically confirmed XLH followed at the Lyon Reference Centre for Rare Calcium, Phosphorus and Magnesium Diseases
* Patients treated with Burosumab
* Patients >12 kg.
* Patients and parent/guardian who have been informed of the study and who do not object to participate

Exclusion Criteria:

* Patients undergoing treatment with oral corticosteroids, or who have received more than 3 months of corticosteroid therapy in the past.
* Patients who have received or are currently receiving immunosuppressive therapy.
* Patients suffering from an inflammatory disease
* Pregnant or breast-feeding women
* Persons deprived of their liberty by judicial or administrative decision
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the Calcium and Phosphate Metabolism Reference Centre:
  * Lyon paediatrics: Femme Mère Enfant hospital (Pr Bacchetta): 20 patients followed
  * Lyon adult section: Edouard Herriot Hospital (Pr S Lemoine, Nephrologist + Dr Vignot, Rheumatologist): 30 patients followed.
    20 patients will be included in the study. The investigators therefore believe that recruitment is fully feasible over 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Expression of inflammatory markers (Il6, Il8, Il1β, CXCL1, CCL2, CXCR3, Il1R, Il6R) obtained from circulating monocytic cells of XLH patients treated with burosumab, before and 7 days after injection. | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Justine Pr BACCHETTA, Pr, Principal Investigator — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No